CLINICAL TRIAL: NCT00912353
Title: A Phase I, Single Center, Randomized, Double-Blind, Placebo-Controlled Single Ascending Oral Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7268 in Healthy Japanese Subjects
Brief Title: AZD7268 Single Ascending Dose Study in Healthy Japanese Subjects
Acronym: JSAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1151C00002
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Phase I; Japanese healthy volunteer; AZD7268

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD7268 (Experimental)
  Interventions: Drug: AZD7268
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7268 — Single Oral
  Arms: AZD7268
Drug: Placebo — Single Oral
  Arms: Placebo

SUMMARY:
This is a Phase I, single center, randomized, double-blind, placebo-controlled single ascending oral dose study to assess the safety, tolerability and pharmacokinetics of AZD7268 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and female (of non-child bearing potential) subjects 20 to 45 years of age, inclusive
* Body weight between 50 and 90 kg, inclusive, with a Body Mass Index (BMI)

  * 18 to ≤ 27 kg/m2

Exclusion Criteria:

* Clinically relevant disease or disorder (past or present), which in the opinion of the investigator, may either put the subject at risk because of participation in the study or influence the results or the subject's ability to participate in the study
* Any clinically significant abnormalities in physical examination, vital signs, clinical chemistry, hematology or urinalysis results as judged by the investigator and/or sponsor
* Smoking in excess of 5 cigarettes per day or equivalent within 30 days of Day 1

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To asses the safety nature and incidence of adverse events, blood pressure, pulse rate, body temperature, physical examination, laboratory assessments (clinical chemistry, hematology, and urinalysis parameters), effects on ECG parameters, EEG recordings, | From screening period to follow-up, 44 days (maiximum).

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD7268 and its metabolite(s) in plasma and urine. | Blood and urine sampling from pre-dose until 72 hrs post dose.
To collect and store DNA for future exploratory research | One blood sampling after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, MD, Principal Investigator — California Clinical Trials
Locations (1):
- Research Site, Gelndale, California, United States